CLINICAL TRIAL: NCT06704750
Title: General Gynecology Center
Brief Title: Correlation Between Physical Fitness Status and Quality of Postoperative Recovery in Gynaecological ERAS Patients
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5257
Record Dates: First submitted 2024-07-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-07

CONDITIONS: Gynecology; Postoperative Recovery; Enhanced Recovery After Surgery; Six-minute Walk Test; EQ5D5L-VAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: 6-minute walk test — patients were instructed to walk back and forth in a marked 30-meter-long straight corridor as fast as they could tolerate
  Other Names: EQ5D5L questionnaire; QOR-15 questiannaire

SUMMARY:
Investigate the current status of perioperative physical fitness.To compare the degree of agreement between the 6-minute walk test and the EQ5D5L-VAS score in assessing recovery after gynecological ERAS, and to provide a reference for a more scientific and comprehensive assessment of patients' physical recovery after gynecological ERAS.

DETAILED DESCRIPTION:
1. Investigate the current status of perioperative physical fitness and postoperative recovery quality of gynaecological ERAS patients
2. Explore the correlation between the physical fitness status of gynaecological ERAS patients and the quality of postoperative recovery.
3. Based on the correlation between patients' physical fitness status and the quality of postoperative recovery, to further determine the optimal threshold of the 6MWT distance

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years old;
* diagnosed with benign gynecological diseases and undergoing laparoscopic surgery;
* acceptance of ERAS modality;
* normal cognitive communication ability and proficiency in the use of smartphones;
* without motor disabilities.

Exclusion Criteria:

* unstable angina and myocardial infarction within 1 month;
* heart rate >120 beats/minute at rest, systolic blood pressure >180 mmHg, diastolic blood pressure >100 mmHg;
* diagnosis of anxiety and depression;
* pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 146 patients were included in this study, and 114 patients completed full follow-up.The average age of the paticipants was 35.48 years old.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | since the preoperative period, followed up until the patients' walk test was fully restored to their follow-up preoperative levels,at most 1 month
  patients were instructed to walk back and forth in a marked 30-meter-long straight corridor as fast as they could tolerate.
EQ5D5L-VAS | since the preoperative period, followed up until the patients' walk test was fully restored to their follow-up preoperative levels, at most 1 month
  5-level EQ-5D version,The first part is a descriptive system, assessing health in five dimensions.The second part of the questionnaire consists of a visual analog scale (VAS) on which patients mark their perceived level of health on a scale ranging from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
QoR-15 | on the preoperative period, on the 1 day of discharge
  15-item Quality of Recovery Scale,the minimum value is 0 and maximum value is 150, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences,Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No